CLINICAL TRIAL: NCT02241291
Title: CARDIOBASE Bern PCI Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 137/14
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Ischemia
Keywords: Percutaneous Coronary Intervention; Registries
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Patients undergoing PCI at Bern University Hospital
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Non-surgical procedure used to treat the stenotic (narrowed) coronary arteries of the heart found in coronary heart disease. A deflated balloon or other device on a catheter is fed from an artery (such as the inguinal femoral artery or radial artery) up through blood vessels until they reach the site of blockage in the heart. X-ray imaging is used to guide the catheter threading. At the blockage, the balloon is inflated to open the artery, allowing blood to flow. A stent is often placed at the site of blockage to permanently open the artery

SUMMARY:
The aim of the CARDIOBASE Bern PCI registry is to collect baseline clinical and procedural data as well as to assess the clinical outcomes of all patients undergoing percutaneous coronary intervention (PCI) at Bern University Hospital. All patients undergoing PCI with or without stent implantation will be prospectively registered. Device use is according to the decision of the treating physician and independent of this registry. At hospital discharge and one year, the following outcomes will be assessed: death, cardiac death, myocardial infarction, stent thrombosis, repeat revascularisation, stent thrombosis, stroke, bleeding, renal failure and vascular complications.

DETAILED DESCRIPTION:
Background

Percutaneous Coronary Intervention (PCI) is the most frequently medical intervention performed worldwide. Coronary heart disease (CAD) remains the leading cause of death, although advances in the management of acute myocardial infarction (MI) have reduced in-hospital mortality from 16% in the mid-1980s to around 4 to 6%. Several breakthroughs have accounted for improvement of cardiovascular outcomes, including the use and further improvement of coronary stents and antiplatelet therapy. Regarding stents, bare metal stents were first introduced but associated with a high risk of restenosis, something which was successfully addressed by the introduction of drug-eluting stents.

All benefits and shortcomings of newly introduced devices and drug therapies are evaluated in large randomized controlled trials (RCT). Registries provide useful insights into novel associations that cannot be addressed by RCT.

The aim of the CARDIOBASE Bern PCI registry is to collect baseline clinical and procedural data as well as to assess the clinical outcomes of all patients undergoing percutaneous coronary intervention at Bern University Hospital. All patients undergoing PCI with or without stent implantation will be prospectively registered. Device use is according to the decision of the treating physician and independent of this registry.

Objective

Prospectively collect baseline clinical, procedural and clinical outcomes at discharge and one year in order to assess the safety and efficacy of PCI at Bern University Hospital.

Methods

ECGs of all patients will be analyzed and a correlation with clinical outcome data performed. Outcomes will be compared in different clinical subgroups. The impact of stent devices implanted and the anti-platelet therapy regimen on cardiovascular outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 years of age
* Undergoing PCI at Bern University Hospital
* Written informed consent

Exclusion Criteria

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective, single-center observational, web-based registry of all patients undergoing percutaneous coronary intervention (PCI) at Bern University Hospital, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-03; Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with death | At discharge, expected to be on average after 2 days, & at one year

SECONDARY OUTCOMES:
Number of patients with myocardial infarction | At discharge, expected to be on average after 2 days, & at one year
Number of patients with stent thrombosis | At discharge, expected to be on average after 2 days, & at one year
Number of patients with repeat revascularisation | At discharge, expected to be on average after 2 days, & at one year
Number of patients with stroke | At discharge, expected to be on average after 2 days, & at one year
Number of patients with bleeding | At discharge, expected to be on average after 2 days, & at one year
Number of patients with | At discharge, expected to be on average after 2 days, & at one year

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, Professor Dr. med., Principal Investigator — Department of Cardiology, Bern University Hospital; Lorenz Raeber, PD Dr. med., Principal Investigator — Department of Cardiology, Bern University Hospital
Locations (1):
- Department of Cardiology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Result] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Result] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Result] Gitt AK, Bueno H, Danchin N, Fox K, Hochadel M, Kearney P, Maggioni AP, Opolski G, Seabra-Gomes R, Weidinger F. The role of cardiac registries in evidence-based medicine. Eur Heart J. 2010 Mar;31(5):525-9. doi: 10.1093/eurheartj/ehp596. Epub 2010 Jan 20. No abstract available. PMID 20093258
- [Result] Mandelzweig L, Battler A, Boyko V, Bueno H, Danchin N, Filippatos G, Gitt A, Hasdai D, Hasin Y, Marrugat J, Van de Werf F, Wallentin L, Behar S; Euro Heart Survey Investigators. The second Euro Heart Survey on acute coronary syndromes: Characteristics, treatment, and outcome of patients with ACS in Europe and the Mediterranean Basin in 2004. Eur Heart J. 2006 Oct;27(19):2285-93. doi: 10.1093/eurheartj/ehl196. Epub 2006 Aug 14. PMID 16908490
- [Derived] Bar S, Kavaliauskaite R, Otsuka T, Ueki Y, Haner J, Lanz J, Furholz M, Praz F, Hunziker L, Siontis GC, Pilgrim T, Stortecky S, Losdat S, Windecker S, Raber L. Quantitative Flow Ratio to Predict Non-Target-Vessel Events Before Planned Staged Percutaneous Coronary Intervention in Patients With Acute Coronary Syndrome. J Am Heart Assoc. 2024 Jan 2;13(1):e031847. doi: 10.1161/JAHA.123.031847. Epub 2023 Dec 29. PMID 38156592
- [Derived] Ueki Y, Zanchin T, Losdat S, Karagiannis A, Otsuka T, Siontis GCM, Haner J, Stortecky S, Pilgrim T, Valgimigli M, Windecker S, Raber L. Self-reported non-adherence to P2Y12 inhibitors in patients undergoing percutaneous coronary intervention: Application of the medication non-adherence academic research consortium classification. PLoS One. 2022 Feb 16;17(2):e0263180. doi: 10.1371/journal.pone.0263180. eCollection 2022. PMID 35171913
- [Derived] Ueki Y, Otsuka T, Bar S, Koskinas KC, Heg D, Haner J, Siontis GCM, Praz F, Hunziker L, Lanz J, Stortecky S, Pilgrim T, Losdat S, Windecker S, Raber L. Frequency and Outcomes of Periprocedural MI in Patients With Chronic Coronary Syndromes Undergoing PCI. J Am Coll Cardiol. 2022 Feb 15;79(6):513-526. doi: 10.1016/j.jacc.2021.11.047. PMID 35144742
- [Derived] Zanchin C, Ledwoch S, Bar S, Ueki Y, Otsuka T, Haner JD, Zanchin T, Praz F, Hunziker L, Stortecky S, Pilgrim T, Losdat S, Windecker S, Raber L, Siontis GCM. Acute coronary syndromes in young patients: Phenotypes, causes and clinical outcomes following percutaneous coronary interventions. Int J Cardiol. 2022 Mar 1;350:1-8. doi: 10.1016/j.ijcard.2022.01.018. Epub 2022 Jan 13. PMID 35033577
- [Derived] Otsuka T, Bar S, Losdat S, Kavaliauskaite R, Ueki Y, Zanchin C, Lanz J, Praz F, Haner J, Siontis GCM, Zanchin T, Stortecky S, Pilgrim T, Windecker S, Raber L. Effect of Timing of Staged Percutaneous Coronary Intervention on Clinical Outcomes in Patients With Acute Coronary Syndromes. J Am Heart Assoc. 2021 Dec 7;10(23):e023129. doi: 10.1161/JAHA.121.023129. Epub 2021 Nov 24. PMID 34816730
- [Derived] Ueki Y, Vogeli B, Karagiannis A, Zanchin T, Zanchin C, Rhyner D, Otsuka T, Praz F, Siontis GCM, Moro C, Stortecky S, Billinger M, Valgimigli M, Pilgrim T, Windecker S, Suter T, Raber L. Ischemia and Bleeding in Cancer Patients Undergoing Percutaneous Coronary Intervention. JACC CardioOncol. 2019 Dec 17;1(2):145-155. doi: 10.1016/j.jaccao.2019.11.001. eCollection 2019 Dec. PMID 34396175
- [Derived] Spirito A, Gragnano F, Corpataux N, Vaisnora L, Galea R, Svab S, Gargiulo G, Siontis GCM, Praz F, Lanz J, Billinger M, Hunziker L, Stortecky S, Pilgrim T, Capodanno D, Urban P, Pocock S, Mehran R, Heg D, Windecker S, Raber L, Valgimigli M. Sex-Based Differences in Bleeding Risk After Percutaneous Coronary Intervention and Implications for the Academic Research Consortium High Bleeding Risk Criteria. J Am Heart Assoc. 2021 Jun 15;10(12):e021965. doi: 10.1161/JAHA.121.021965. Epub 2021 Jun 8. PMID 34098740
- [Derived] Ueki Y, Bar S, Losdat S, Otsuka T, Zanchin C, Zanchin T, Gragnano F, Gargiulo G, Siontis GCM, Praz F, Lanz J, Hunziker L, Stortecky S, Pilgrim T, Heg D, Valgimigli M, Windecker S, Raber L. Validation of the Academic Research Consortium for High Bleeding Risk (ARC-HBR) criteria in patients undergoing percutaneous coronary intervention and comparison with contemporary bleeding risk scores. EuroIntervention. 2020 Aug 28;16(5):371-379. doi: 10.4244/EIJ-D-20-00052. PMID 32065586
- [Derived] Zanchin C, Ueki Y, Zanchin T, Haner J, Otsuka T, Stortecky S, Koskinas KC, Siontis GCM, Praz F, Moschovitis A, Hunziker L, Valgimigli M, Pilgrim T, Heg D, Windecker S, Raber L. Everolimus-Eluting Biodegradable Polymer Versus Everolimus-Eluting Durable Polymer Stent for Coronary Revascularization in Routine Clinical Practice. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1665-1675. doi: 10.1016/j.jcin.2019.04.046. Epub 2019 Aug 14. PMID 31422088
- [Derived] Ueki Y, Karagiannis A, Zanchin C, Zanchin T, Stortecky S, Koskinas KC, Siontis GCM, Praz F, Otsuka T, Hunziker L, Heg D, Moschovitis A, Seiler C, Billinger M, Pilgrim T, Valgimigli M, Windecker S, Raber L. Validation of High-Risk Features for Stent-Related Ischemic Events as Endorsed by the 2017 DAPT Guidelines. JACC Cardiovasc Interv. 2019 May 13;12(9):820-830. doi: 10.1016/j.jcin.2018.12.005. Epub 2019 Apr 10. PMID 30981574
- [Derived] Yamaji K, Zanchin T, Zanchin C, Stortecky S, Koskinas KC, Hunziker L, Praz F, Blochlinger S, Moro C, Moschovitis A, Seiler C, Valgimigli M, Billinger M, Pilgrim T, Heg D, Windecker S, Raber L. Unselected Use of Ultrathin Strut Biodegradable Polymer Sirolimus-Eluting Stent Versus Durable Polymer Everolimus-Eluting Stent for Coronary Revascularization. Circ Cardiovasc Interv. 2018 Sep;11(9):e006741. doi: 10.1161/CIRCINTERVENTIONS.118.006741. PMID 30354590
- [Derived] Li J, Wyrsch D, Heg D, Stoller M, Zanchin T, Perrin T, Windecker S, Raber L, Roten L. Electrocardiographic predictors of mortality in patients after percutaneous coronary interventions - a nested case-control study. Acta Cardiol. 2019 Aug;74(4):341-349. doi: 10.1080/00015385.2018.1494117. Epub 2018 Oct 17. PMID 30328801
- [Derived] Zanchin T, Temperli F, Karagiannis A, Zanchin C, Rasanen M, Koskinas KC, Stortecky S, Hunziker L, Praz F, Blochlinger S, Moro C, Moschovitis A, Seiler C, Billinger M, Heg D, Pilgrim T, Valgimigli M, Windecker S, Raber L. Frequency, Reasons, and Impact of Premature Ticagrelor Discontinuation in Patients Undergoing Coronary Revascularization in Routine Clinical Practice: Results From the Bern Percutaneous Coronary Intervention Registry. Circ Cardiovasc Interv. 2018 May;11(5):e006132. doi: 10.1161/CIRCINTERVENTIONS.117.006132. PMID 29748219
- [Derived] Koskinas KC, Zanchin T, Klingenberg R, Gencer B, Temperli F, Baumbach A, Roffi M, Moschovitis A, Muller O, Tuller D, Stortecky S, Mach F, Luscher TF, Matter CM, Pilgrim T, Heg D, Windecker S, Raber L. Incidence, Predictors, and Clinical Impact of Early Prasugrel Cessation in Patients With ST-Elevation Myocardial Infarction. J Am Heart Assoc. 2018 Apr 13;7(8):e008085. doi: 10.1161/JAHA.117.008085. PMID 29654204
- [Derived] Zanchin T, Raber L, Koskinas KC, Piccolo R, Juni P, Pilgrim T, Stortecky S, Khattab AA, Wenaweser P, Bloechlinger S, Moschovitis A, Frenk A, Moro C, Meier B, Fiedler GM, Heg D, Windecker S. Preprocedural High-Sensitivity Cardiac Troponin T and Clinical Outcomes in Patients With Stable Coronary Artery Disease Undergoing Elective Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2016 Jun;9(6):e003202. doi: 10.1161/CIRCINTERVENTIONS.115.003202. PMID 27296200
- [Derived] Koskinas KC, Raber L, Zanchin T, Wenaweser P, Stortecky S, Moschovitis A, Khattab AA, Pilgrim T, Blochlinger S, Moro C, Juni P, Meier B, Heg D, Windecker S. Clinical impact of gastrointestinal bleeding in patients undergoing percutaneous coronary interventions. Circ Cardiovasc Interv. 2015 May;8(5):e002053. doi: 10.1161/CIRCINTERVENTIONS.114.002053. PMID 25910501